CLINICAL TRIAL: NCT01218009
Title: A Multi-Center 52-Week Study to Assess the Safety of an Albuterol Dry-powder Inhaler in Subjects With Asthma
Brief Title: A Twelve Month Long Term Safety Study to Evaluate the Safety of Albuterol in a Dry Powder Inhaler With Both Repeated and as Needed Dosing
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change to study required.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-306
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
Keywords: asthma; dry powder inhaler; short-acting beta2-agonist; SABA; bronchoconstriction; bronchodilation; bronchodilator; metered dose inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol Spiromax (Experimental): Albuterol multi-dose dry powder inhaler (Spiromax) at a dose of 720 micrograms per day administered as 2 inhalations of 90 mcg /inhalation four times a day for the 12 week double-blind period. Participants then continue into the 40 week open-label period in which they take albuterol multi-dose dry powder inhaler (Spiromax) inhalations of 90 mcg /inhalation as required (PRN).
  Interventions: Drug: Albuterol Spiromax
- Placebo Spiromax (Placebo Comparator): Placebo delivered using a multi-dose dry powder inhaler (Spiromax) as 2 inhalations four times a day for the 12 week double-blind period. Participants then continue into the 40 week open-label period in which they administer albuterol multi-dose dry powder inhaler (Spiromax) inhalations of 90 mcg /inhalation as required (PRN).
  Interventions: Drug: Placebo Spiromax; Drug: Albuterol Spiromax

INTERVENTIONS:
Drug: Placebo Spiromax — Placebo as a dry-powder inhaled orally using the Spiromax inhaler. During the 12-week double-blind period, participants take two (2) inhalations four times a day (QID) at approximately 7:00 AM, 12:00 PM, 5:00 PM, and bedtime.
  Arms: Placebo Spiromax
Drug: Albuterol Spiromax — Albuterol as a dry-powder inhaled orally using the Spiromax inhaler. Each inhalation delivers 90 micrograms (mcg). During the 12-week double-blind period, participants take two (2) inhalations four times a day (QID) at approximately 7:00 AM, 12:00 PM, 5:00 PM, and bedtime for a total dose of 720 micrograms per day for those paricipants randomized to the Albuterol treatment arm.
  The double-blind period is followed by a 40-week open-label period in which all study participants will take Albuterol Spiromax 90 micrograms (mcg)/inhalation as needed (PRN).
  Other Names: ProAir® RespiClick, Albuterol multi-dose dry powder inhaler (MDPI)

SUMMARY:
This is a one-year study to look at the safety of a dry powder inhaler with albuterol. After a one-week run in, for the first 3 months subjects will use an inhaler with either albuterol or a dummy drug at regular times four times a day. Then for the last nine months of the study, all subjects will be given the albuterol dry powder inhaler and will use it only when needed to help with breathing problems. Subjects will need to keep a daily diary (both paper and electronic) throughout the study recording any inhaler use and health problems. There will be visits to the study doctor about once a month for a year. This study is intended to show that the albuterol dry powder inhaler works well and is safe for use over a long period of time.

DETAILED DESCRIPTION:
The Sponsor terminated this study due to the need for a modification to the Spiromax device utilized in this study; the problem identified has no impact on patient safety. Exposure ranged from 3 to 49 days with the majority of subjects receiving ≤30 days of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of persistent asthma with rescue use of albuterol on average of at least once/ week over the 4-weeks prior to screening.
* Female subjects who are of childbearing potential (as judged by the investigator) must be currently using and willing to continue to use a medically reliable method of contraception for the entire study duration
* General good health
* Capable of understanding the requirements, risks, and benefits of study participation
* Non-smoker for at least one year prior to the screening visit and a maximum pack-year smoking history of 10 years
* Other criteria apply

Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study related visit
* Participation in any investigational drug trial within 30 days preceding the screening visit
* A known hypersensitivity to albuterol or any of the excipients in the formulations.
* History of severe milk protein allergy
* History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, otitis media, influenza, etc) which is not resolved within 1 week prior to the Screening Visit.
* Use of any protocol prohibited concomitant medications for asthma or any protocol prohibited concomitant non-asthma medications
* Inability to tolerate or unwillingness to comply with the protocol requirements.
* History of life-threatening asthma
* Any asthma exacerbation within 3 months of the Screening Visit requiring oral or systemic corticosteroids
* History of life-threatening asthma
* Other criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Teva Respiratory R&D
Locations (30):
- United States (30):
  - Teva Clinical Study Site, Scottsdale, Arizona
  - Teva Clinical Study Site, Los Angeles, California
  - Teva Clinical Study Site, San Diego, California
  - Teva Clinical Study Site, Centennial, Colorado
  - Teva Clinical Study Site, Denver, Colorado
  - Teva Clinical Study Site, Miami, Florida
  - Teva Clinical Study Site, Gainesville, Georgia
  - Teva Clinical Study Site, Louisville, Kentucky
  - Teva Clinical Study Site, Wheaton, Maryland
  - Teva Clinical Study Site, Minneapolis, Minnesota
  - Teva Clinical Study Site, Plymouth, Minnesota
  - Teva Clinical Study Site, St Louis, Missouri
  - Teva Clinical Study Site, Bellevue, Nebraska
  - Teva Clinical Study Site, Boys Town, Nebraska
  - Teva Clinical Study Site, Skillman, New Jersey
  - Teva Clinical Study Site, Rochester, New York
  - Teva Clinical Study Site, Rockville Centre, New York
  - Teva Clinical Study Site, High Point, North Carolina
  - Teva Clinical Study Site, Raleigh, North Carolina
  - Teva Clinical Study Site, Canton, Ohio
  - Teva Clinical Study Site, Cincinnati, Ohio
  - Teva Clinical Study Site, Sylvania, Ohio
  - Teva Clinical Study Site, Eugene, Oregon
  - Teva Clinical Study Site, Portland, Oregon
  - Teva Clinical Study Site, El Paso, Texas
  - Teva Clinical Study Site, New Braunfels, Texas
  - Teva Clinical Study Site, San Antonio, Texas
  - Teva Clinical Study Site, Burke, Virginia
  - Teva Clinical Study Site, Seattle, Washington
  - Teva Clinical Study Site, Greenfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four hundred fifty-two patients were screened and 331 randomized into the study.
Period: Overall Study
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Started | 166 | 165
Completed | 0 | 0
Not Completed | 166 | 165
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Sponsor terminated study | 161 | 163

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol Spiromax | Placebo Spiromax | Total
Number analyzed (Participants) | 166 | 165 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.07) | 38.0 (14.91) | 37.9 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 122 | 227
  Male | 61 | 43 | 104
Race/Ethnicity, Customized [Number; unit: participants]
  White | 140 | 132 | 272
  Black | 19 | 28 | 47
  Asian | 4 | 1 | 5
  North American or Alaska Native | 1 | 0 | 1
  Other | 2 | 4 | 6
Ethnicity [Number; unit: participants]
  Hispanic | 20 | 21 | 41
  Not Hispanic | 146 | 144 | 290
Height [Mean (Standard Deviation); unit: inches] | 66.1 (3.59) | 65.7 (3.86) | 65.9 (3.73)
Weight [Mean (Standard Deviation); unit: pounds] | 184 (49.7) | 179 (48.2) | 182 (48.9)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Day 49 (study termination)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 166 | 165
participants
  Any adverse event | 59 | 58
  Treatment-related adverse event | 3 | 3
  Withdrawn from study due to adverse event | 0 | 0
  Serious adverse event | 1 | 1
  Treatment-related serious adverse event | 0 | 0
  Mild adverse event | 29 | 32
  Moderate adverse event | 35 | 29
  Severe adverse event | 2 | 4
  AE class: Infections and infestations | 31 | 34
  AE class: Respiratory, thoracic and mediastinal | 12 | 11
  AE class: Gastrointestinal | 9 | 5
  AE class: Nervous system | 7 | 6
  AE class: Injury, poisoning and procedural compli | 4 | 2
  AE class: Investigations | 3 | 3
  AE class: Musculoskeletal and connective tissue | 2 | 4
  AE class: Renal and urinary | 2 | 1
  AE class: Ear and labyrinth | 2 | 1
  AE class: Skin and subcutaneous tissue | 2 | 0
  AE class: General and administrative site conditi | 1 | 1
  AE class: Psychiatric | 1 | 1
  AE class: Social circumstances | 1 | 0
  AE class: Cardiac | 0 | 2
  AE class: Eye | 0 | 1
  AE class: Blood and lymphatic system | 0 | 1
  Neoplasm benign, malignant + unspecified | 0 | 1

2. Primary Outcome: Changes From Screening in the Results of the Physical Examination That Are Clinically Significant in the Opinion of the Investigator
Description: A complete physical examination was planned at study screening, week 12 and week 52 or early termination/discontinuation of the participant. At weeks 12 and 52,the qualified healthcare professional was to evaluate whether each physical finding is a new finding, worsening, improvement or resolution of an existing condition compared with the baseline physical exam. Where possible, the same qualified healthcare professional that performed the physical examination at study screening should perform all the scheduled physical examinations.
Time Frame: Days -15 to -8 (Screening), Week 12, Week 52
Population: Safety population. The study was terminated prior to the during study evaluations.
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Changes From Screening in the Results of the Laboratory Evaluations That Are Clinically Significant in the Opinion of the Investigator
Description: Blood samples were to collected for laboratory evaluations at the screening visit and at weeks 12 and 52 or early termination/discontinuation of the participant. The blood samples were to be drawn after an overnight fast of at least 6 hours and analyzed by a central laboratory.
Time Frame: Days -15 to -8 (Screening), Week 12, Week 52
Population: Safety population. The study was terminated prior to the during study evaluations.
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Changes From Screening in the Results of the Electrocardiograms (ECGs) That Are Clinically Significant in the Opinion of the Investigator
Description: A standard 12-lead ECG was to be performed at screening and at week 12 and week 52 (TV15) or early termination/discontinuation of the participant. The ECG recording methods were to be centralized and standardized across all study subjects.
Time Frame: Days -15 to -8 (Screening), Week 12, Week 52
Population: Safety population. The study was terminated prior to the during study evaluations.
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Changes From Screening in the Vital Signs That Are Clinically Significant in the Opinion of the Investigator
Description: Vital sign measurements (heart rate and blood pressure) were to be evaluated as part of the safety profile assessment. The participant was to be seated at least 2 minutes before vital signs were performed. Either an electronic or manual sphygmomanometer could be used.
Time Frame: Days -15 to -8 (Screening), Week 12, Week 52
Population: Safety population. The study was terminated prior to the during study evaluations.
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 0 | 0

6. Post Hoc Outcome: Blood Pressure at Screening and End of Study
Description: Vital sign measurements (heart rate and blood pressure) were evaluated as part of the safety profile assessment. The participant was seated at least 2 minutes before vital signs were performed. Either an electronic or manual sphygmomanometer was used.
Time Frame: Days -15 to -8 (Screening), up to Day 49 (End of study)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 166 | 165
mmHg
  Screening Diastolic BP (n=166, 165) | 75.5 (9.24) | 75.2 (9.08)
  End of Study Diastolic BP (n=164, 164) | 75.7 (9.54) | 75.2 (8.79)
  Screening Systolic BP (n=166, 165) | 119.4 (13.39) | 118.0 (13.70)
  End of Study Systolic BP (n=164, 164) | 118.4 (13.50) | 118.2 (12.99)

7. Post Hoc Outcome: Pulse at Screening and End of Study
Description: Vital sign measurements (heart rate and blood pressure) were evaluated as part of the safety profile assessment. The participant was seated at least 2 minutes before vital signs were performed. Heart rate was measured by radial pulse.
Time Frame: Days -15 to -8 (Screening), up to Day 49 (End of study)
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Number analyzed (Participants) | 166 | 165
beats/minute
  Screening (n=166, 165) | 71.0 (8.57) | 71.8 (10.03)
  End of study (n=164, 164) | 72.1 (9.34) | 73.0 (9.48)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 49 (study termination)
Arm/Group | Albuterol Spiromax | Placebo Spiromax
Serious Adverse Events (participants affected / at risk) | 1/166 | 1/165
Other Adverse Events (participants affected / at risk) | 16/166 | 20/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol Spiromax (N=166) | Placebo Spiromax (N=165)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol Spiromax (N=166) | Placebo Spiromax (N=165)
Nasopharyngitis (Infections and infestations) | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data